CLINICAL TRIAL: NCT01720771
Title: Preventive Effect of a Probiotic Tablet on Oral Health in Preschool Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Svante Twetman, Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EPN-2011/530; EPN-2011/530 (Other: Etikprovningsnamnden)
Record Dates: First submitted 2012-10-31; First posted 2012-11-02 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Dental Caries
Keywords: bacteriotherapy; caries; preschool children; probiotics
MeSH Terms: conditions — Dental Caries | interventions — Probiotics; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic tablet (Active Comparator): a tablet with three probiotic streptococci strains (S. uberis KJ2, S. oralis KJ3 and S. rattus JH145) at a concentration of 3x108 CFU
  Interventions: Dietary Supplement: probiotic tablet
- Sugar pill (Placebo Comparator): The same tablet but without active probiotic bacteria
  Interventions: Dietary Supplement: sugar pill

INTERVENTIONS:
Dietary Supplement: probiotic tablet — Intake of one probiotic lozenge tablet per day
  Other Names: Evora Kids
  Arms: Probiotic tablet
Dietary Supplement: sugar pill — one tablet daily
  Other Names: Evora kids (placebo)
  Arms: Sugar pill

SUMMARY:
The aim of the prospective project is to investigate effect of daily probiotic supplements on dental caries development in preschool children living in a low socioeconomic immigrant area in souithern Sweden. The study design is a randomised controlled trial with two parallell arms. The intervention is one probiotic tablet or placebo once daily. The null hypothesis is that the caries experience and increment will not differ betwwen the two groups.

DETAILED DESCRIPTION:
Background In spite of the general decline in dental caries, early childhood caries (ECC) is still a severe global problem with social and behavioural gradients [1, 2]. The disease is multi-factorial but the key event is a pH-induced stress in the oral environment that results in reduced diversity of the oral biofilm [3]. The biofilm simply adapt to this situation with an overgrowth of caries-associated aciduric strains on behalf of beneficial and health promoting bacteria. Therefore, the addition of probiotic bacteria has been suggested as a novel approach to maintain oral health as an adjunct to the existing evidence-based methods [4, 5]. Previous clinical trials have indicated that a daily intake of lactobacilli-derived dairy products can reduce caries incidence, improve general health and diminish the use of antibiotics in preschool children [6, 7, 8]. However, further studies on the probiotic concept are needed; all children do not drink milk and no studies on childhood caries have hitherto been conducted with non-dairy products and streptococci strains.

Objectives The aim of the present project is to evaluate the effect of daily administration of chewing tablets containing probiotic bacteria (Probiora3) on plaque amount, gingival health and caries incidence in preschool children. In addition, information on general health will be collected. The null hypothesis is that the oral health will not differ from preschool children with a similar intake of placebo tablets. An additional aim is to monitor the microbial composition in saliva samples at baseline and during the course of intervention.

Study design The study design is a prospective randomised, double-blind, placebo-controlled trial with two parallel arms. The duration is 12 months. Assignment to intervention and control group will be made by a computer-based randomization in groups A or B.

Material The study group will be recruited among the 2-year-old children that are regular patients attending the Public Dental Clinic in Rosengård, Malmö, Sweden. The clinic is situated in a multicultural suburban area with a low socio-economy. The proportion of immigrants is high in the area, the majority Arabic speaking. The inclusion criteria are i) uncompromised general health, ii) no cavities or severe dental diseases, and iii) not mentally or physically disabled. Children that are uncooperative or totally reject dental examination are excluded. The children will be consecutively enrolled after signed informed consent (verbal and written) by their parents and assigned to either the test or the control group by pre-numbered envelopes generated by a computer program. As a new patient is entering the study, the clinician takes the next numbered envelope assigning the patient to either group A or B. The protocol has been subjected to the regional ethical committee and is approved.

Power calculation A power calculation of the clinical scores with alpha set at 0.05 and beta = 0.2 estimates that 85 subjects in each arm is needed to disclose a 30% difference between the treatment groups with respect to the clinical scores (Fleiss Statistical Methods for rates and Proportions, 2nd edition, John Wiley and Sons New York 1981). Due to expected relocations and failure to comply with the protocol, the goal will be to recruit a minimum of 220 and a maximum of 250 children.

Intervention and duration All families will receive comprehensive reinforcement of the oral health message by their dental hygienists prior to baseline. The focus will be on daily supervised brushing with fluoride toothpaste. At the baseline examination, plaque index, bleeding after brushing and caries are scored on special forms for optical reading. Data on ongoing medication etc will be extracted from the dental records. In addition, a caries risk assessment is carried out with the aid of a computerized program (Cariogram) according to Stecksén-Blicks et al. 2007 [8]. The parents of the children in the test-group (group A) will be instructed to give their children one EvoraKids® tablet once daily, ideally after brushing, for a period of 12 months. The parents of the children in the control-group (group B) will receive the same instructions for the intake of tablets without live probiotic bacteria. The group assignment will be unknown both for the parents and the investigators and disclosed only after the statistical calculations. The allocation concealment is kept by the manufacturer. All parents are encouraged to maintain all their habitual oral hygiene routines and use fluoride toothpaste throughout the study period.

The test tablets contain Probiora3 which is a trade mark for three probiotic streptococci strains (S. uberis KJ2, S. oralis KJ3 and S. rattus JH145) at a concentration of 3x108 CFU. The tablets are sweetened by erythritrol which is a tooth-friendly polyol (for nutrition facts, see Appendix B). The chew tablets (test and placebo), identical in taste and appearance, will be supplied by the manufacturer (Oragenics, USA) in packages separated by the letter "A" or "B". The participating families will be provided with tablets for three month's use at the time and the compliance will be checked and registered at each follow-up. Parents will be instructed to report any perceived side- or adverse-effects immediately to the dental staffs and stop the intake.

Clinical examinations

Clinical examinations will be performed at baseline and after 6 and 12 months. The families are contacted every third month for interviews and delivery of study products. The examinations and scoring will be carried out visually and tactile by two well-trained and calibrated dental hygienists at the dental clinic. At baseline, information on the domestic oral hygiene routines, use of baby bottles and habitual sweet dietary intakes will be collected by a 10-question questionnaire. The following endpoints are scored:

Primary outcome measures:

* visible plaque index (VPI)
* prevalence of gingival inflammation (bleeding after brushing, BAB)
* prevalence of caries (cavitated lesions and white spot lesions)

Secondary outcome measures:

* number of upper or lower respiratory infections
* number of otitis media
* number of days with diarrhea
* doctor's visits
* prescription of antibiotics
* incidence of allergy, asthma or eczema

Detailed methodology Visible plaque index (VPI): Presence or absence of dental plaque along the gingival margin of the upper incisors and canines Bleeding after brushing (BAB): Presence/absence of bleeding after gentle brushing with a soft toothbrush Presence of caries: Cavitated and non-cavitated lesions are registered in all teeth according to the criterion of the Public Dental Service and expressed as dmft and dmfs

The secondary endpoints are scored every sixth month through telephone calls to the parents and based on parental logbooks.

Clinical sampling In order to monitor the oral microbiota in the 2 study groups during the course of the study, saliva samples will be collected at baseline (before intervention) and at the 6 and 12 months follow-ups according to Barfod and co-workers [9]. A cotton bud is placed by the parents in the mouth of their child under supervision of the clinical staff. When soaked, the bud will be transferred to a small plastic tube, marked with the patients study number, and immediately frozen and stored. After the full completion of the trial, all samples will be shipped on expense of the manufacturer to Oragenics, FL, USA for further handling and processing. The running costs for the clinical samplings are covered by a separate agreement.

Statistical methods All data are processed with the IBM-SPSS software (version 19.0, Chicago IL, USA). The categorical data are subjected chi-square tests. Continuous measurements will be calculated with aid of non-parametric tests. The caries incidence is calculated as the difference in dmfs/dmft between follow-up and baseline. Comparisons are carried out between the study groups at baseline and at the follow-ups. The group concealment will not be unveiled until after the statistical calculations. A p value less than 0.05 is considered as statistically significant.

Report of results The null hypothesis will either be rejected or accepted. The findings will without any unnecessary delay be reported at an international congress and submitted for publication to an appropriate peer-reviewed scientific journal. The suppliers will have a the possibility to read and comment on the manuscript before submission.

Ethical considerations There are no side- or adverse-effects to be foreseen in connection with the intervention. All the patients are managed by dentists or specially trained dental hygienists according to "best clinical practice" during and after the project. A rapid development of caries will be managed by non-operative and operative treatment irrespective of group. All treatment will be carried out without costs for the families. The tablets are distributed free of charge. All adverse events related to the treatment provided will be recorded on an adverse event form. The investigation will be performed according to the principles of the Declaration of Helsinki on experimentation involving human subjects.

ELIGIBILITY:
Inclusion Criteria:)

* uncompromised general health,
* no cavities or severe dental diseases,
* and not mentally or physically disabled

Exclusion Criteria:

* Children that are uncooperative or totally reject dental examination are excluded

Ages: 2 Years to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 138 (Actual)
Dates: Start 2013-02; Primary Completion 2014-12 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Caries increment in primary teeth | after 1 year of intervention
  Caries is recorded by clinical examinations with mirror and explorer

CONTACTS AND LOCATIONS:
Locations (1):
- Public Dental Clinic, Folktandvården Rosengård, Wachtmeistersväg 13, Malmo, Skåne County, Sweden

REFERENCES:
- [Derived] Hedayati-Hajikand T, Lundberg U, Eldh C, Twetman S. Effect of probiotic chewing tablets on early childhood caries--a randomized controlled trial. BMC Oral Health. 2015 Sep 24;15(1):112. doi: 10.1186/s12903-015-0096-5. PMID 26403472